CLINICAL TRIAL: NCT06361069
Title: The Efﬁcacy of Finger Puppets, Distraction Cards and Kaleidoscope for Reducing Anxiety in Children Undergoing Day Surgery
Brief Title: Reducing Anxiety in Children Undergoing Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Aslı Akdeniz Kudubeş, ASSOCIATE PROFESSOR, Bilecik Seyh Edebali Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: aslıakdeniz
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Child, Only; Surgery
Keywords: Anxiety; Child; Day surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was conducted using the "pre-post test unpaired group model", one of the quasi-experimental methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 20 children in the control group
- Experimental group (Experimental): 22 in the finger puppet, 21 in the distraction cards intervention group, and 22 in the kaleidoscope intervention group
  Interventions: Other: distraction cards, kaleidoscope and finger puppet

INTERVENTIONS:
Other: distraction cards, kaleidoscope and finger puppet — A kaleidoscope, characterized by vibrant patterns visible through rotation of its cylinders, operates on the principle of light refraction, producing dynamic and ever-changing visual displays.
  Distraction cards feature an array of images and shapes, each measuring approximately 5-8 cm in length. These intricate designs are discernible only upon careful examination of the cards.
  Puppets, as a therapeutic intervention tool, significantly influence children's personal, social, and emotional development, facilitating their comfortable expression of emotions.
  Arms: Experimental group

SUMMARY:
Aim: This study was conducted to determine the efﬁcacy of finger puppets, distraction cards and kaleidoscope for reducing anxiety in children undergoing day surgery.

Methods: The study was conducted using the "pre-post test unmatched group model", one of the quasi-experimental methods. The study was conducted between April 2023 and January 2024 with children aged 6-12 years who were admitted to the pediatric clinic of a hospital for day surgery. A total of 85 children (including 20 children in the control group, 22 children in the finger puppet intervention group, 21 children in the distraction cards intervention group, and 22 children in the kaleidoscope intervention group) who were hospitalized in the pediatric clinic between April 2023 and January 2024 and who met the inclusion criteria were included in the study. Descriptive statistics, Mann Whitney U test, Kruskal Wallis and regression analysis were used in the evaluation of the data.

DETAILED DESCRIPTION:
This study was conducted to determine the efﬁcacy of finger puppets, distraction cards and kaleidoscope for reducing anxiety in children undergoing day surgery. The study was conducted using the "pre-post test unpaired group model", one of the quasi-experimental methods.

The study was carried out from April 2023 to January 2024, involving children aged 6-12 years admitted to the pediatric clinic of a teaching and research hospital for day surgery (tonsillectomy, circumcisio, adenotonsillectomy etc.). Notably, the nursing care provided at the hospital does not incorporate distraction techniques aimed at alleviating anxiety in children.

Sample The sample required for the study was calculated using the G*Power (3.1.9.4) computer program. Based on the Type I error of 5%, Type II error of 99%, SD = 6.20, and Type I error of 5% in the study by Dehghan et al. (2017), the desired effect size for this study was 0.55 and the total required sample size was 64 children (approximately 21 children for each group) (Dehghan et al., 2017). A total of 85 children, comprising 20 children in the control group, 22 in the finger puppet intervention group, 21 in the distraction cards intervention group, and 22 in the kaleidoscope intervention group, was recruited from the pediatric clinic between April 2023 and January 2024, meeting the study's inclusion criteria. Notably, no randomization method was employed in the selection process.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-12 years
* scheduled for day surgery
* devoid of prior surgical experiences
* willingly consented to participation.

Exclusion Criteria:

* children undergoing major surgeries (e.g., cardiac procedures)
* emergency surgical interventions
* individuals with mental retardation
* as well as those with visual or auditory impairments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | up to 10 months
  This study was conducted to determine the efﬁcacy of finger puppets, distraction cards and kaleidoscope for reducing anxiety in children undergoing day surgery

CONTACTS AND LOCATIONS:
Overall Officials: ASLI AKDENİZ KUDUBEŞ, phd, Principal Investigator — BİLECİK ŞEYH EDEBALİ UNIVERSITY
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No